CLINICAL TRIAL: NCT05648643
Title: Arterial Elastance: A Predictor of Hypotension Due to Anesthesia Induction
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Serap Aktaş, Medical doctor, Acibadem University
Other Study IDs: ATADEK 2021-10/21
Record Dates: First submitted 2022-11-26; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Hemodynamic Instability; Anesthesia
Keywords: General anesthesia; Arterial elastance; Post-induction hypotension; Monitorization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypotension is very common during and after anesthesia induction. A prolonged fasting period, a patient's underlying comorbidities, a sympathetic blockade by anesthetic agents, vasodilation, a reduction in preload, and cardiac contractility can cause post-induction hypotension.1,2 The relationship of even short-term hypotension with myocardial damage, renal injury, and stroke has been shown in many studies; therefore, it is very important to provide stable anesthesia induction.3 In current anesthesia practice, we can only intervene when hypotension occurs. If we can identify patients who may experience hypotension during anesthesia induction before it occurs, we can prevent possible postoperative organ dysfunctions by reducing the duration and depth of hypotension with prophylactic fluid and vasopressor administration. We hypothesized that arterial elastance (Ea) values before anesthesia induction could predict post-induction hypotension. To test our hypothesis, we aimed to investigate the reliability of the Ea value, which was monitored preoperatively using the pressure analytical recording method (PRAM) to predict the risk of hypotension that may occur after anesthesia induction.

DETAILED DESCRIPTION:
Anesthesia induction-related hypotension is not uncommon and is still challenging for anesthesiologists to predict, despite advanced monitoring techniques. In current anesthesia practices, approximately 20-30% of patients develop hypotension during and after anesthesia induction. In large observational studies, the relationship between intraoperative hypotension and adverse cardiac, renal, and cerebral outcomes has been reported. Approximately one-third of intraoperative hypotension episodes occur during and after the induction of anesthesia, and most can be prevented if foreseeable. Therefore, we need quick and easy markers to predict patients at risk of hypotension to achieve the stable induction of anesthesia.

Many studies have used noninvasive and invasive monitoring techniques for the preoperative prediction of hypotension after anesthesia induction.

However, most studies evaluate the cardiovascular system with parameters that determine the preload and fluid responsiveness to predict the risk of post-induction hypotension, though the arterial system and its interaction with the ventricle are ignored.The heart and the arterial system are both anatomically and functionally interconnected and do not act independently. The major determinant of cardiovascular system performance and cardiac energetics is ventriculoarterial coupling (VAC). Ea is an indicator of cardiac afterload and arterial tone and can be calculated by the ratio of the end-systolic pressure (ESP) and stroke volume (SV) obtained from arterial wave analysis.Ea provides information about the ESP/SV relationship and dynamic afterload and gives the clinician the opportunity to evaluate VAC indirectly. We hypothesized that Ea values before anesthesia induction could predict post-induction hypotension. To test our hypothesis, we aimed to investigate the reliability of the Ea value, which was monitored preoperatively using the pressure analytical recording method (PRAM) to predict the risk of hypotension that may occur after anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA( American Society Of Anesthesiology) physical status 1-3
* Underwent major elective surgery
* Required intra-arterial blood pressure monitoring before induction.

Exclusion Criteria:

* Under 18 years of age
* Arrhythmia (atrial fibrillation, frequent premature beat)
* Severe pre-existing lung disease
* Severe valvular heart disease
* morbid obesity
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with ASA physical status 1-3 who underwent major elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Arterial elastance (Ea) measured before anesthesia induction was investigated whether is a predictive parameter for post-induction hypotension in patients undergoing general anesthesia. | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Ea ((mmHg m-2ml-1)is an indicator of cardiac afterload and arterial tone and can be calculated by the ratio of the end-systolic pressure (ESP) and stroke volume (SV) obtained from arterial wave analysis. Ea was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy) before the anesthesia induction

SECONDARY OUTCOMES:
Stroke volume variation (SVV), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Stroke volume variation (SVV,%), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). SVV is a parameter used to asses cardiac preload and fluid responsiveness

OTHER OUTCOMES:
Pulse pressure variation (PPV), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Pulse pressure variation (PPV,%) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). PPV is a parameter used to asses cardiac preload and fluid responsiveness.
Cardiac power output (CPO), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Cardiac power output (CPO, Watt) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). CPO is a parameter used to asses cardiac reserve
Cardiac index (CI), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Cardiac index (CI, L/min/m2), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). CI is a parameter used to asses cardiac stroke volume
Dp/Dt, measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Dp/Dt(mmHg/msn), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). Dp/Dt is a parameter used to asses cardiac contractility.
Systolic arterial pressure (SAP), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Systolic arterial pressure (SAP- mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). SAP is a parameter used to assess the pressure of the arterial system during cardiac systole
diastolic arterial pressure (DAP), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Diastolic arterial pressure (DAP, mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). DAP is a parameter used to assess the pressure of the arterial system during cardiac diastole.
mean arterial pressure (MAP), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Mean arterial pressure (MAP, mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). MAP is a parameter used to assess organ perfusion.
Heart rate (HR), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Heart rate (HR/bpm) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). HR is a parameter used to assess the cardiac rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monge Garcia MI, Jian Z, Settels JJ, Hatib F, Cecconi M, Pinsky MR. Reliability of effective arterial elastance using peripheral arterial pressure as surrogate for left ventricular end-systolic pressure. J Clin Monit Comput. 2019 Oct;33(5):803-813. doi: 10.1007/s10877-018-0236-y. Epub 2018 Dec 14. PMID 30552525
- [Background] Merillon JP, Ennezat PV, Guiomard A, Masquet-Gourgon C, Aumont MC, Gourgon R. Left ventricular performance is closely related to the physical properties of the arterial system: Landmark clinical investigations in the 1970s and 1980s. Arch Cardiovasc Dis. 2014 Oct;107(10):554-62. doi: 10.1016/j.acvd.2014.08.001. Epub 2014 Oct 8. PMID 25304173
- [Background] Monge Garcia MI, Jian Z, Settels JJ, Hunley C, Cecconi M, Hatib F, Pinsky MR. Determinants of left ventricular ejection fraction and a novel method to improve its assessment of myocardial contractility. Ann Intensive Care. 2019 Apr 16;9(1):48. doi: 10.1186/s13613-019-0526-7. PMID 30993544